CLINICAL TRIAL: NCT04414982
Title: An Intervention to Increase Engagement With Hypertension Care for American Indian Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Heart Association (Other); University of Colorado Centers for American Indian and Alaska Native Health (Unknown); Denver Health and Hospital Authority (Other); Denver Indian Health and Family Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 15-1711
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Hypertension
Keywords: Hypertension; Medication Adherence; Values Affirmation; American Indian/Alaska Native
MeSH Terms: conditions — Hypertension; Medication Adherence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Values Affirmation (Experimental): Compare the effects of the values-affirmation exercise with a control exercise in AI/AN patients with hypertension.
  Interventions: Behavioral: Intervention Values Affirmation
- Control Values Affirmation (Active Comparator): Compare the effects of the values-affirmation exercise in AI/AN patients with its effects in white patients.
  Interventions: Behavioral: Control Values Affirmation

INTERVENTIONS:
Behavioral: Intervention Values Affirmation — Participants are asked to circle the two or three values that are MOST important to them. Next, participants are asked to think about times when the values chosen might be important to THEMSELVES and then write a few sentences to describe when and why they might be important.
  Arms: Intervention Values Affirmation
Behavioral: Control Values Affirmation — Participants are asked to circle the two or three items that are LEAST important to them. Next, participants are asked to think about times when the values chosen might be important to SOMEONE ELSE and then write a few sentences to describe when and why they might be important.
  Arms: Control Values Affirmation

SUMMARY:
The objective of this study is to reduce the effects of stereotype threat on the adherence of American Indian/Alaska Native patients with hypertension.

The specific aims of this study, which employs a values affirmation intervention, are to:

1. Compare the effects of the values-affirmation exercise with a control exercise in AI/AN patients with hypertension.
2. Compare the effects of the values-affirmation exercise in AI/AN patients with its effects in white patients.

DETAILED DESCRIPTION:
American Indians and Alaska Natives (AI/ANs) in the U.S. bear a disproportionate burden of cardiovascular disease. They have a higher prevalence of conditions that predispose to cardiovascular disease and poorer outcomes after developing cardiovascular disease than white Americans. The causes of these differences are complex and multiple, but there are widespread concerns that racial bias contributes to the problem. As concluded over a decade ago in the 2003 Institute of Medicine report, Unequal Treatment, "Racial/ethnic disparities in health care occur in the context of broader historic and contemporary social and economic inequality and evidence of persistent racial and ethnic discrimination… Bias, stereotyping and prejudice on the part of healthcare providers may contribute to racial and ethnic disparities in health care." These concerns persist. Minority group members are well aware of negative stereotypes targeted at them as a group and of the possibility of bias directed at them as individuals. Given the reality of prejudice and their previous experiences with it, it is understandable that minority group members would be apprehensive about the possibility of being judged in light of the stereotype, both outside and inside the healthcare system. Critically, this apprehension may occur in the absence of actual bias. This raises the possibility that interventions directed at patients' perception of discrimination may have an independent and additive effect beyond the effects of interventions directed at provider bias.

Investigators propose to evaluate a novel intervention that reduces the detrimental effects of negative stereotypes on minority patients by reducing stereotype threat through values- affirmation. Stereotype threat is a stressful psychological state that occurs when a person fears being judged in light of negative stereotypes. The stress of this situation and the pressure to avoid confirming negative stereotypes can result in impaired performance and worse outcomes - something of a self-fulfilling prophecy. For example, an American Indian patient fearful of confirming the stereotype of being unintelligent may fail to ask for clarification of changes in antihypertensive medications and, based on misconceptions, persist in taking an old regimen that is ineffective. Values-affirmation is a process in which global sense of personal worth is strengthened in the face of a threat, making individuals better able to cope with psychological threats.

The intervention proposed in this application is based on one found to be effective in alleviating stereotype threat in other contexts such as education and in alleviating more general threats to the self in a health context as well as in a prior study investigators performed with African American patients. Investigators will randomly assign AI/AN patients with hypertension to complete an affirmation exercise or a control exercise prior to a visit with their providers. The affirmation exercise is performed immediately before a clinic visit. It asks patients to reflect on values or self-defining skills that they find important, and to write a few sentences about why one of them is important. The project is innovative in that it is directed against a mechanism, stereotype threat, not generally recognized as important in healthcare settings. Since the intervention is brief and easily applied across a wide range of health conditions, it directly addresses the need for interventions to be generalizable and sustainable.

ELIGIBILITY:
Inclusion Criteria:

* Hypertension diagnosis: primary or secondary ICD-10 code diagnosis in last 24 mo
* SBP >160 mm Hg or DBP >90 mm Hg in last 12 months
* Currently taking antihypertensive medications
* Medications filled within health system's pharmacy
* White or American Indian/Alaska Native, self-reported race
* Upcoming primary care visit
* Ability to read and write English
* History of hypertension defined as having an outpatient visit in the past year with a primary or secondary ICD-9 code diagnosis of hypertension, with the diagnosis of hypertension confirmed by review of the patient's medical record before enrollment.
* Additional inclusion criteria are age >18 years
* Use of Denver Indian Health and Family Services (DIHFS) or Denver Health (DH) as their usual source of care.
* American Indian/Alaska Native as defined by DIHFS uses to define eligibility for no-cost services.
* To define the comparator group at DH we will use self-described race/ethnicity of white/non- Latino.
* All eligible patients must have the ability to provide informed consent.

Exclusion Criteria:

* Pregnancy-related hypertension
* Dialysis-dependent end-stage renal disease
* Patients who cannot speak or write English
* Unable to provide consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Change in Antihypertensive Medication Adherence using Pharmacy Records | Baseline, 3 and 6 months
  This antihypertensive medication adherence outcome will be a summary measure of adherence which assesses the proportion of days covered (PDC) over the period of observation for which a patient obtains antihypertensive medications. Adherence will be calculated for each antihypertensive drug in the regimen and combined across drugs into a summary measure of adherence for the entire drug regimen.
Change in Antihypertensive Medication Adherence using Self-Reported Adherence | Baseline, 3 and 6 months
  This antihypertensive medication adherence outcome will be a summary measure of self-reported adherence using the validated Voils instrument, which has 3 questions that address adherence over the previous 7 days.
Change in Antihypertensive Medication Adherence using Pill Counts | Baseline, 3 and 6 months
  This antihypertensive medication adherence outcome will be a summary outcome measure of adherence where if x is the number of pills in the bottle, y is the number of pills that would have been in the bottle had all pills been taken since the bottle was filled, and z is the number of pills that should have been taken since the last fill, and adherence is calculated as 1- [(x-y)/z].

SECONDARY OUTCOMES:
Systolic Blood Pressure | Baseline, 3 and 6 months
  Systolic blood pressure over time.
Proportion of Time Blood Pressure is Under Control | 6 months
  Defined as the proportion of time over the 6-months of follow-up with a BP ≤ 160/90 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Ed Havranek, MD, Principal Investigator — University of Colorad, Denver
Locations (2):
- United States (2):
  - Denver Health and Hospital Authority, Denver, Colorado
  - Denver Indian Health and Family Services, Denver, Colorado

REFERENCES:
- [Derived] Gust CJ, Bryan AD, Havranek EP, Vupputuri S, Steiner JF, Blair IV, Hanratty R, Daugherty SL. Health Behavior Theory and Hypertension Management: Comparisons Among Black, White, and American Indian and Alaska Native Patients. Race Soc Probl. 2022 Dec;14(4):369-382. doi: 10.1007/s12552-022-09359-2. Epub 2022 Feb 25. PMID 38322707